CLINICAL TRIAL: NCT05907369
Title: Disgust Reduction Through Evaluative Conditioning and tDCS in Patients With Contamination-Based OCD
Brief Title: Disgust Reduction Through Evaluative Conditioning (DREC) and tDCS in Contamination-Based OCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ferdowsi University of Mashhad (Other)
Responsible Party: Principal Investigator, Ali Moghimi, Professor, Ferdowsi University of Mashhad
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 3/56765; 100/18979 (Other: Cognitive Sciences and Technologies Council of Iran)
Record Dates: First submitted 2023-05-15; First posted 2023-06-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Contamination symptoms; Disgust; Evaluative Conditioning; Transcranial Direct Current Stimulation; Orbitofrontal Cortex
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: The two interventions include evaluative conditioning (EC) training and cathodal tDCS over OFC. Each is present in two forms: active and sham. So, there are four interventional conditions, including sham EC-sham tDCS, active EC- sham tDCS, sham EC-active tDCS, and active EC-active tDCS.
Who Masked: Participant
Masking Description: Participants are blind to which of the interventions is active or a sham. Interventional sessions look the same for all participants regarding duration and activities (including doing a computerized EC task and receiving tDCS).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- aEC/ stDCS (Experimental): Participants in this group receive active EC training but sham tDCS.
  Interventions: Other: Active EC training; Other: Sham tDCS
- sEC/atDCS (Active Comparator): Participants in this group receive active tDCS training but sham EC training.
  Interventions: Other: Sham EC training; Other: Active tDCS
- aEC/atDCS (Experimental): Participants in this group receive both active EC training and active tDCS.
  Interventions: Other: Active EC training; Other: Active tDCS
- sEC/stDCS (Sham Comparator): Participants in this group receive the sham EC training and also sham tDCS.
  Interventions: Other: Sham EC training; Other: Sham tDCS

INTERVENTIONS:
Other: Active EC training — The active EC includes pairing contamination-related pictures (CSs) with pleasant pictures (USs). The EC training takes about 15 minutes and is administered for ten sessions (5 days a week) in 4 difficulty levels.
  Arms: aEC/ stDCS; aEC/atDCS
Other: Sham EC training — The active EC includes pairing contamination-related pictures (CSs) with neutral pictures (USs). The EC training takes about 15 minutes and is administered for ten sessions (5 days a week) in 4 difficulty levels, the same as active EC training.
  Arms: sEC/atDCS; sEC/stDCS
Other: Active tDCS — For the active tDCS, the cathode is placed over the left OFC and the anode over the right cerebellum. The brain stimulation is delivered with a 2mA current intensity for 20 minutes in 10 sessions (5 days a week).
  Arms: aEC/atDCS; sEC/atDCS
Other: Sham tDCS — For the sham tDCS, the cathode is placed over the left OFC and the anode over the right cerebellum, the same as active tDCS. The device is on for 20 minutes, but the current intensity is under the threshold of affecting cortical activity modulation. The participants receive the sham tDCS in 10 sessions (5 days a week).
  Arms: aEC/ stDCS; sEC/stDCS

SUMMARY:
Obsessive-compulsive disorder (OCD) is a debilitating health condition that is known by intrusive and unwanted thoughts and repetitive behavioral or mental acts. 2-3% of the population suffers from OCD in their lifetime. The most common OCD subtype is contamination. The Serotonin-selective reuptake inhibitors (SSRIs) and cognitive-behavioral therapy (CBT) based on exposure and response prevention (ERP) technique are the first-line treatments for OCD. The challenge is that nearly half do not respond to the first-line treatments or have residual symptoms after completion of treatments. However, the prevalence of the disorder, diversity of symptoms, inadequate response rate, and necessity of having long-lasting treatment effects make the treatments of OCD more challenging.

It seems that abnormal, more intense disgust experience has a prominent role in developing and maintaining OCD symptoms, particularly the contamination subtype. Evaluative conditioning (EC), defined as transferring the value of the US to the CS through pairing them, is the most common way of establishing disgust responses. The present study aims to develop an emotion-based intervention technique using EC targeting disgust emotion in contamination-based OCD (C-OCD). The hypothesis is that EC training may modify disgust experiences. Disgust may be the culprit, at least in part, of cognitive deficiencies in OCD. The other hypothesis is whether disgust reduction-focused EC may improve cognitive function, such as attention bias and inhibitory control.

The orbitofrontal cortex (OFC) is one of the brain areas engaged in disgust processing and is mostly hyperactive in OCD patients. Cathodal transcranial direct current stimulation (tDCS) over OFC is one of the helpful neuromodulation methods in treating OCD. We aim to see if this method may help to regulate disgust experiences in combination with EC. The participants may be referred by psychiatrists or psychotherapists or be self-referred due to online advertisements or paper flyers. They will be randomly assigned to one of for arms of the study for sham or active EC training along with sham or active tDCS, to which they are blind. The novelty of the present study is the application of EC training in the clinical OCD population in combination with a neuromodulation method.

DETAILED DESCRIPTION:
Disgust as a primary emotion has evolved to protect our lives by driving dirt and disease avoidance behaviors and motivating for cleaning and hygienic behaviors. In recent years, many studies have focused on the role of disgust in psychiatric disorders such as anxiety disorders, eating disorders, body dysmorphic disorders, and phobias. Nowadays, we have robust evidence of the correlation between disgust and the etiology and treatment of OCD symptoms, particularly the contamination subtype. The principal explanation for the insufficient treatment effect of ERP is that disgust is resistant to extinction.

Since evaluative conditioning is one of the main sources of disgust feeling, the same process may effectively reduce disgust. The present trial will try to pair contamination-related pictures that are disgust-eliciting with positive, pleasant pictures in order to modify their disgust valence. We also will administer this EC training plus to OFC cathodal tDCS to see if the EC effect becomes more significant than EC alone.

ELIGIBILITY:
Inclusion Criteria:

* The Diagnostic criteria of OCD in the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5-TR) with the symptoms of contamination subtype
* Able to read, write and do computerized tasks
* Stable medication for at least the last three months
* Filling out the written consent

Exclusion Criteria:

* Severe physical illness
* Severe other mental disorders
* Alcohol and drug dependence
* A history of epilepsy or seizure
* Have metal or electronic implants in the head or use a cardiac pacemaker
* History of head trauma or neurological disorders
* Women who are pregnant or may be pregnant
* Unable to complete questionnaires, computerized tasks, or informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
Disgust Feeling | From pre- to post-assessment (2 weeks after baseline assessment) and from pre- to follow-up assessment (10 weeks after baseline assessment)
  Effect of evaluative conditioning, cathodal tDCS over OFC, and both on changing disgust feeling intensity measured by disgust rating scale. The scale rates from 0 (not disgusting) to 10 (very disgusting). Lower scores show less disgust feeling.
Clinical Symptoms Severity of Contamination-Based OCD | From pre- to post-assessment (2 weeks after baseline assessment) and from pre- to follow-up assessment (10 weeks after baseline assessment)
  Change in Clinical symptoms of contamination-based OCD after evaluative conditioning, cathodal tDCS over OFC, and both, measured by Yale-Brown Obsessive-Compulsive scale. It is scored on a 5-point rating. The lower scores show less symptom severity.

SECONDARY OUTCOMES:
The power spectrum of brain waves based on quantitative electroencephalogram | From pre- to post-assessment (2 weeks after baseline assessment) and from pre- to follow-up assessment (10 weeks after baseline assessment)
  Effect of evaluative conditioning, cathodal tDCS over OFC, and both on power spectrum of recorded brain waves.
Attentional bias | From pre- to post-assessment (2 weeks after baseline assessment) and from pre- to follow-up assessment (10 weeks after baseline assessment)
  Change in attentional bias toward contamination stimuli, measured by Dot-prob test, comparing evaluative conditioning, cathodal tDCS over OFC, and both.
Inhibitory control | From pre- to post-assessment (2 weeks after baseline assessment) and from pre- to follow-up assessment (10 weeks after baseline assessment)
  Change in inhibitory control, measured by go/nogo and stop-signal tests, comparing evaluative conditioning, cathodal tDCS over OFC, and both.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Moghimi, PhD, Study Director — Ferdowsi University of Mashhad
Locations (1):
- Ferdowsi University of Mashhad, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Mohaddesin FR, Moghimi A, Fadardi JS. Disgust-reduction evaluative conditioning (DREC) and brain stimulation in patients with contamination-based obsessive-compulsive disorder: a protocol for a randomized control trial. Trials. 2023 Nov 24;24(1):750. doi: 10.1186/s13063-023-07791-2. PMID 38001473